CLINICAL TRIAL: NCT01897636
Title: Efficacy and Safety of Endoscopic Ultrasound Guided Fine-needle Injection of Dendritic Cells Vaccination Into Unresectable Pancreatic Cancer
Acronym: DC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Ying Lv, Associate professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zkx12019
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Cancer
Keywords: endoscopic ultrasound-guided fine-needle injection; dendritic cell; vaccination
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUS-guided fine-needle injection of DCs vaccinations (Experimental)
  Interventions: Procedure: EUS-guided fine-needle injection of DCs vaccinations

INTERVENTIONS:
Procedure: EUS-guided fine-needle injection of DCs vaccinations

SUMMARY:
Pancreatic cancer is the second most frequent gastrointestinal malignancy. The overall survival is dismal. Especially for advanced pancreatic cancer, the conventional approaches are typically not curative and provide only minor increases in survivals in most cases. Dendritic cells (DCs) are powerful antigen-presenting cells (APCs) that play a pivotal role in the initiation, programming, and regulation of tumor-specific immune responses. Isolated DCs loaded with tumor antigen ex vivo and administered as a cellular vaccine have been found to induce protective and therapeutic anti-tumor immunity in experimental animals. Some clinical trials of DC vaccination for cancer patients have shown the induction of anti-tumor immune responses and tumor regression. Endoscopic ultrasound (EUS) is an established technique for the diagnosis and staging of pancreatic cancer. Endoscopic ultrasound guided fine-needle direct injection of dendritic cells vaccination into pancreatic tumors may be a promising treatment modality.Therefore, The purpose of the study is to evaluate the efficacy and safety of endoscopic ultrasound guided fine-needle injection of DCs vaccination into advanced pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas.
2. Patients must be deemed unresectable due to involvement of important vasculature, adjacent organ invasion, presence of metastasis, or other medical condition making surgical resection unfavorable.
3. Life expectancy of >3 months.
4. Karnofsky performance status >50%.
5. Patients must have adequate clotting and coagulation function (platelet > 100k; INR<1.4).
6. Able and willing to sign a written informed consent.

Exclusion Criteria:

1. Patients receiving anticoagulation therapy.
2. Steroids or immunosuppressing agent dependant status
3. Patients who have received prior gemcitabine or radiation therapy in the past 4 weeks
4. Ongoing infection
5. Pregnancy or breast-feeder
6. Other concurrent diseases including other malignancy,psychiatric illness,heart, lung and renal disfunctions
7. Massive ascites
8. Decision of unsuitableness by principal investigator or physician-in-charge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
pancreatic tumor response rates | six months

SECONDARY OUTCOMES:
survival rates | six month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Zou, PhD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum-Tower Hospital, Nanjing, Jiangsu, China